CLINICAL TRIAL: NCT05969067
Title: Comparing Retroperitoneal Tunneling Versus Dissection Technique During Robotic Assisted Sacrocolpopexy for Pelvic Organ Prolapse
Brief Title: Retroperitoneal Tunneling Versus Dissection Technique During Sacrocolpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0124
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Sacrocolpopexy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dissection Technique (Placebo Comparator): The peritoneum is incised superficially and opened longitudinally from the sacral promontory, downward to the posterior cul-de-sac and the posterior vaginal wall to create retroperitoneal space for the SCP mesh.
  Interventions: Procedure: Dissection Technique during RA SCP
- Tunneling Technique (Experimental): A retroperitoneal tunnel is created by undermining the peritoneum with the robotic scissors and/or needle driver which is placed in the peritoneal opening over the sacral promontory. The tunnel is created just medial to the right uterosacral ligament and toward the posterior vaginal wall by using forward pressure and a sweeping motion to create a space within the retroperitoneum
  Interventions: Procedure: Tunneling Technique during RA SCP

INTERVENTIONS:
Procedure: Tunneling Technique during RA SCP — As described in the intervention arm above
  Arms: Tunneling Technique
Procedure: Dissection Technique during RA SCP — As described in the intervention arm above
  Arms: Dissection Technique

SUMMARY:
The purpose of this study is to compare operative time, patient reported outcomes, surgical complications, and surgical outcomes between the tunneling versus dissection technique during robotic assisted sacrocolpopexy (RA SCP).

DETAILED DESCRIPTION:
Women with symptomatic, stage II to IV POP who plan RA SCP at UTMB Health will be approached to participate. Using the study protocol inclusion and exclusion criteria, patient's eligibility will be determined. All eligible subjects will provide the written informed consent before any research data is collected. All screening assessments will be completed at a preoperative, in-person, clinic visit, and within 60 days of surgery. The subject will then undergo randomization to tunneling versus dissection technique during RA SCP with the total sample size of 40 female subjects (20 per group). Concomitant procedures for POP or urinary incontinence are permitted and will be based upon the operating surgeons' standard clinical practice and best clinical judgement. Subsequently, the subject will have postoperative follow up at 2 weeks, 6 weeks and 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Females at least 18 years of age at the time of consent.
2. Able to understand and read English
3. Able and willing to provide written informed consent
4. Able to comply with the follow-up study protocol, per clinician judgment
5. Symptomatic POP (bulge or pressure) evidenced with vaginal prolapse with POP-Q measurement consistent with Stage II-IV.
6. RA SCP as desired surgical approach to correct apical prolapse

Exclusion Criteria:

1. Females who are pregnant, or intend to become pregnant during the study
2. Texas Department of Criminal Justice prisoners
3. A known history of sensitivity to propylene mesh
4. Prior prolapse repair surgery using mesh (abdominal, vaginal or rectal)
5. Active or chronic systemic infection including any pelvic infection, abscess
6. Has had history of primary pelvic organ cancer (uterine, ovarian, endometrial, cervical, bladder) or any cancer that is metastatic to the pelvis
7. Prior or current pelvic radiation, or chemotherapy.
8. Not a candidate for general anesthesia
9. History of systemic connective tissue or musculoskeletal disorders (scleroderma, SLE, Marfan's syndrome, Ehlers Danlos, polymyositis, Lambert Eaton syndrome etc)
10. History of neurologic condition affecting bladder function (multiple sclerosis, spinal cord injury, stroke with neurologic deficit)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Operative Time (minutes) | Intraoperative time
  Operating time for dissection technique: includes dissection and suturing time. The dissection time starts when the robotic instruments are used to extend the retroperitoneal incision (created during the presacral space dissection) and ends when the extension reaches the posterior vaginal wall. The suturing time starts when the needle enters the peritoneum at the presacral space and ends when the suture is cut after the presacral space, retroperitoneal space and the peritoneum covering the mesh are completely re-approximated.
  Operating time for tunneling technique: includes tunneling and suturing time. The tunneling time starts when the robotic instruments are used to undermine the peritoneum and ends when the tunnel is completely created, reaching the posterior vaginal wall. The suturing time starts when the needle enters the peritoneum to close the presacral space and ends when the suture is cut after the peritoneum covering the mesh is completely re-approximated.

SECONDARY OUTCOMES:
POP-Q exam | Baseline, 6 weeks postoperatively and 12 weeks postoperatively
  The POP-Q is staged by using the 9 measurements. The stage can range from good support (no organ descent) reported as a POP-Q stage 0 or I to a POP-Q score of IV (complete procidentia or vault eversion)
Pelvic Floor Distress Inventory PFDI-20 | Baseline, 6 weeks postoperatively and 12 weeks postoperatively
  The questionnaire is scored from 0-300. Higher scores indicate being worse (more distressing)
Pelvic Floor Impact Questionnaire PFIQ-7 | Baseline, 6 weeks postoperatively and 12 weeks postoperatively
  The questionnaire is scored from 0-300. Higher scores indicate being worse (more distressing)
Pelvic Organ Prolapse/ Urinary Incontinence Sexual Questionnaire PISQ-12 | Baseline, 6 weeks postoperatively and 12 weeks postoperatively
  The total score of the PISQ-12 questionnaire ranges from 0 to 48. The higher the score is, the better the quality of sexual life.
Patient Global Impression of Improvement PGI-I | Baseline, 6 weeks postoperatively and 12 weeks postoperatively
  Report the patient's response using the response scale from 1-7
Decision Regret Scale (DRS) | 6 weeks postoperatively and 12 weeks postoperatively
  A five-item paper and pencil self-report measure that asks subjects to reflect on a particular decision and then rate each item on a Likert scale from 1 (strongly agree) to 5 (strongly disagree). Higher scores are worse.
Satisfaction with Decision Scale (SDS) | 6 weeks postoperatively and 12 weeks postoperatively
  Scoring consists of taking the mean of the 6 items (range 1 to 5)
Clavien-Dindo classification for operative complication | 2 weeks, 6 weeks postoperatively and 12 weeks postoperatively
  The system is used to grade adverse events related to surgical procedures from 1 to 5. Higher grade indicates worse adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Kilic, MD, Principal Investigator — UTMB
Locations (1):
- University of Texas Medical Branch Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers

REFERENCES:
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Maher C, Feiner B, Baessler K, Christmann-Schmid C, Haya N, Brown J. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2016 Oct 1;10(10):CD012376. doi: 10.1002/14651858.CD012376. PMID 27696355
- [Background] Paraiso MFR, Jelovsek JE, Frick A, Chen CCG, Barber MD. Laparoscopic compared with robotic sacrocolpopexy for vaginal prolapse: a randomized controlled trial. Obstet Gynecol. 2011 Nov;118(5):1005-1013. doi: 10.1097/AOG.0b013e318231537c. PMID 21979458
- [Background] Erekson EA, Yip SO, Ciarleglio MM, Fried TR. Postoperative complications after gynecologic surgery. Obstet Gynecol. 2011 Oct;118(4):785-93. doi: 10.1097/AOG.0b013e31822dac5d. PMID 21934441
- [Background] Kim EK, Applebaum JC, Kravitz ES, Hinkle SN, Koelper NC, Andy UU, Harvie HS. "Every minute counts": association between operative time and post-operative complications for patients undergoing minimally invasive sacrocolpopexy. Int Urogynecol J. 2023 Jan;34(1):263-270. doi: 10.1007/s00192-022-05412-1. Epub 2022 Nov 23. PMID 36418567
- [Background] Hoshino K, Yoshimura K, Nishimura K, Hachisuga T. How to reduce the operative time of laparoscopic sacrocolpopexy? Gynecol Minim Invasive Ther. 2017 Jan-Mar;6(1):17-19. doi: 10.1016/j.gmit.2016.05.005. Epub 2016 Jul 5. PMID 30254863
- [Background] Guan X, Ma Y, Gisseman J, Kleithermes C, Liu J. Robotic Single-Site Sacrocolpopexy Using Barbed Suture Anchoring and Peritoneal Tunneling Technique: Tips and Tricks. J Minim Invasive Gynecol. 2017 Jan 1;24(1):12-13. doi: 10.1016/j.jmig.2016.06.012. Epub 2016 Jun 23. PMID 27344033
- [Background] Liu J, Bardawil E, Zurawin RK, Wu J, Fu H, Orejuela F, Guan X. Robotic Single-Site Sacrocolpopexy with Retroperitoneal Tunneling. JSLS. 2018 Jul-Sep;22(3):e2018.00009. doi: 10.4293/JSLS.2018.00009. PMID 30356342
- [Background] Pushkar DY, Kasyan GR, Popov AA. Robotic sacrocolpopexy in pelvic organ prolapse: a review of current literature. Curr Opin Urol. 2021 Nov 1;31(6):531-536. doi: 10.1097/MOU.0000000000000932. PMID 34506336
- [Background] Matanes E, Boulus S, Lauterbach R, Amit A, Weiner Z, Lowenstein L. Robotic laparoendoscopic single-site compared with robotic multi-port sacrocolpopexy for apical compartment prolapse. Am J Obstet Gynecol. 2020 Apr;222(4):358.e1-358.e11. doi: 10.1016/j.ajog.2019.09.048. Epub 2019 Oct 4. PMID 31589864
- [Background] Halder GE, White AB, Brown HW, Caldwell L, Wright ML, Giles DL, Heisler CA, Bilagi D, Rogers RG. A telehealth intervention to increase patient preparedness for surgery: a randomized trial. Int Urogynecol J. 2022 Jan;33(1):85-93. doi: 10.1007/s00192-021-04831-w. Epub 2021 May 24. PMID 34028575

DOCUMENTS (1):
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT05969067/ICF_000.pdf